CLINICAL TRIAL: NCT02727686
Title: Post-Operative Water Load Following Transsphenoidal Pituitary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Barrow Brain and Spine (Unknown); Barrow Neurological Institute (Other)
Responsible Party: Principal Investigator, Pam Dewey, Research Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PHX1600103012
Record Dates: First submitted 2016-03-23; First posted 2016-04-05 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Hyponatremia; Pituitary Adenoma
Keywords: transsphenoidal pituitary surgery
MeSH Terms: conditions — Hyponatremia; Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Water Load (WL) Post-Operative Day 1 (Experimental): All enrolled subjects passing conditions outlined in Intervention are eligible to be included. WL will be calculated (20 mL/kg body weight) and supplied at the bedside. Patient will have 30 minutes to consume WL, or will be excluded.
  Interventions: Other: Water Load (WL) Post-Operative Day 1

INTERVENTIONS:
Other: Water Load (WL) Post-Operative Day 1 — Patient will have normonatremic 0600 hr sodium level (Serum Sodium = 135 - 145 mmol/L), ability to safely take water by mouth, and cleared to continue by treating surgeon. WL will be calculated (20 mL/kg body weight) and supplied at the bedside. Vasopressin level will be determined. Patient will have 30 minutes to consume WL, or will be excluded. Included patients will have data collected as follows: 1 hour - serum sodium, urine output; 2 hour - serum sodium, urine output, vasopressin level; 6 hours - serum sodium, urine output.

SUMMARY:
Delayed post-operative hyponatremia occurs in 5-20% of patients following pituitary surgery and typically occurs on post-operative day 5-10.This decline in sodium can occur rapidly and have serious consequences such as altered mental status, seizures, coma, and even death. Despite significant research into patient demographics and risk factors, the investigators have not been able to predict which patients will suffer from delayed post-operative hyponatremia to date. At the Barrow Neurological Institute, physicians currently utilize an outpatient screening protocol to monitor patients' sodium levels after surgery, but this has yet to be effective for reducing readmissions following pituitary surgery. The etiology of delayed post-operative hyponatremia has been linked to water and sodium dysregulation in the post-operative period. It has been shown that post-operative day 1-2 sodium levels are statistically lower in patients who develop delayed hyponatremia, however, the numerical differences are not large enough to guide clinical management. The investigators propose that a water load on post-operative day 1 may expose underlying sodium/water dysregulation in the early post-operative period. This would improve physicians' understanding of the pathophysiology of post-operative hyponatremia, and it may help to serve as a screening tool for these patients in the future.

DETAILED DESCRIPTION:
Current standards are for screening of all post-operative transsphenoidal pituitary patients for sodium abnormalities in the POD(post-operative day)7-14 window. At the Barrow Neurological Institute, physicians have instituted a universal screening protocol for all post-operative patients wherein all patients have a serum sodium level drawn on POD5-7 and attempts are made to manage mild to moderate hyponatremia on an outpatient basis.This screening protocol has effectively identified delayed post-operative hyponatremia, however, it has yet to reduce readmissions for hyponatremia in these patients. The researchers propose that implementing a water load test on POD1 may facilitate outpatient screening in three ways: 1) The water load may identify a subset of patients who have appropriate water and sodium regulation after surgery and do not require close monitoring of outpatient sodium levels. 2) The water load may identify a subset of patients who are at risk for delayed hyponatremia and would benefit from strict counseling and closer outpatient monitoring. 3) The water load may identify a subset of patients with a moderate to severe reduction in serum sodium in response to the water load, and these patients may benefit from further monitoring in the hospital prior to discharge. If any of these scenarios hold true, this may change the way physicians monitor and treat patients following transsphenoidal surgery in the future. Furthermore, this protocol could be readily expanded to other neurosurgery practices and could facilitate care for future patients undergoing transsphenoidal pituitary surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Functioning or non-functioning pituitary adenoma
* Sodium level 135-145 prior to surgery

Exclusion Criteria:

* Enrolled in a separate pituitary research study
* Unable to provide his/her own consent
* Unable to take PO water
* Renal insufficiency
* Require maintenance corticosteroids pre-operatively
* TSH secreting tumor
* Patients who the treating surgeon deems a poor candidate for the water challenge
* Prisoners
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
POD1 Response Serum Sodium | Post-Operative Day 1
  Evaluate patients' responses to water load on the morning of post-operative day 1: serum sodium (normal range 135-145 mmol/L)
POD1 Response Serum Osmolality | Post-Operative Day 1
  Evaluate patients' responses to water load on the morning of post-operative day 1: serum osmolality (normal range 275-300 mOsm/kg)
POD1 Response Urine Output | Post-Operative Day 1
  Evaluate patients' responses to water load on the morning of post-operative day 1: urine output (normal range > 0.5 ml/kg/hr)
POD1 Response Vasopressin | Post-Operative Day 1
  Evaluate patients' responses to water load on the morning of post-operative day 1: vasopressin level (normal range 0.0 - 6.9 pg/ml)

SECONDARY OUTCOMES:
Post-Discharge Response | Post-Operative Day 2-7
  Follow patients' serum sodium levels after discharge from the hospital and assess for any correlation in water load response and outpatient sodium levels. This is not done with a mathematical calculation but by observation of lab results. Hypothetically, normal water load response (serum sodium =135-145) will equate to normal outpatient sodium levels (135-145). Likewise, an abnormal water load response (sodium < 135 or >145) will equate to possible abnormal outpatient sodium levels (< 135, >145).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Little, MD, Principal Investigator — Barrow Brain and Spine, Phoenix AZ
Locations (1):
- Barrow Brain and Spine, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussain NS, Piper M, Ludlam WG, Ludlam WH, Fuller CJ, Mayberg MR. Delayed postoperative hyponatremia after transsphenoidal surgery: prevalence and associated factors. J Neurosurg. 2013 Dec;119(6):1453-60. doi: 10.3171/2013.8.JNS13411. Epub 2013 Sep 20. PMID 24053496
- [Background] Bohl MA, Ahmad S, Jahnke H, Shepherd D, Knecht L, White WL, Little AS. Delayed Hyponatremia Is the Most Common Cause of 30-Day Unplanned Readmission After Transsphenoidal Surgery for Pituitary Tumors. Neurosurgery. 2016 Jan;78(1):84-90. doi: 10.1227/NEU.0000000000001003. PMID 26348011
- [Background] Olson BR, Gumowski J, Rubino D, Oldfield EH. Pathophysiology of hyponatremia after transsphenoidal pituitary surgery. J Neurosurg. 1997 Oct;87(4):499-507. doi: 10.3171/jns.1997.87.4.0499. PMID 9322839
- [Background] Kristof RA, Rother M, Neuloh G, Klingmuller D. Incidence, clinical manifestations, and course of water and electrolyte metabolism disturbances following transsphenoidal pituitary adenoma surgery: a prospective observational study. J Neurosurg. 2009 Sep;111(3):555-62. doi: 10.3171/2008.9.JNS08191. PMID 19199508
- [Background] Taylor SL, Tyrrell JB, Wilson CB. Delayed onset of hyponatremia after transsphenoidal surgery for pituitary adenomas. Neurosurgery. 1995 Oct;37(4):649-53; discussion 653-4. doi: 10.1227/00006123-199510000-00007. PMID 8559292
- [Background] Chen L, White WL, Spetzler RF, Xu B. A prospective study of nonfunctioning pituitary adenomas: presentation, management, and clinical outcome. J Neurooncol. 2011 Mar;102(1):129-38. doi: 10.1007/s11060-010-0302-x. Epub 2010 Aug 21. PMID 20730474
- [Background] Zada G, Liu CY, Fishback D, Singer PA, Weiss MH. Recognition and management of delayed hyponatremia following transsphenoidal pituitary surgery. J Neurosurg. 2007 Jan;106(1):66-71. doi: 10.3171/jns.2007.106.1.66. PMID 17236489
- [Background] Staiger RD, Sarnthein J, Wiesli P, Schmid C, Bernays RL. Prognostic factors for impaired plasma sodium homeostasis after transsphenoidal surgery. Br J Neurosurg. 2013 Feb;27(1):63-8. doi: 10.3109/02688697.2012.714013. Epub 2012 Aug 21. PMID 22905890
- [Background] Kelly DF, Laws ER Jr, Fossett D. Delayed hyponatremia after transsphenoidal surgery for pituitary adenoma. Report of nine cases. J Neurosurg. 1995 Aug;83(2):363-7. doi: 10.3171/jns.1995.83.2.0363. PMID 7616287